CLINICAL TRIAL: NCT00759668
Title: Visual Function and Patient Satisfaction After Bilateral Implantation of AcrySof Natural ReSTOR (Model SN60D3) or AcrySof Natural Monofocal (Model SN60AT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Marcello Fornoni, Alcon
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IT 06 01
Record Dates: First submitted 2008-09-24; First posted 2008-09-25 (Estimated); Results first posted 2011-01-26 (Estimated); Last update posted 2011-01-26 (Estimated); Status verified 2011-01

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SN60D3 (Experimental): AcrySof Natural ReSTOR Intraocular Lens (IOL) Model SN60D3
  Interventions: Device: Acrysof Natural ReSTOR SN60D3
- SN60AT (Active Comparator): AcrySof Natural Monofocal Intraocular Lens (IOL) Model SN60AT
  Interventions: Device: Acrysof Natural Monofocal SN60AT

INTERVENTIONS:
Device: Acrysof Natural ReSTOR SN60D3 — Bilateral implantation with the AcrySof Natural ReSTOR Intraocular Lens (IOL) SN60D3 following cataract removal.
  Arms: SN60D3
Device: Acrysof Natural Monofocal SN60AT — Bilateral implantation with the AcrySof Natural Intraocular Lens (IOL) Model SN60AT following cataract removal.
  Arms: SN60AT

SUMMARY:
The purpose of the study is:

* to compare visual parameters (Subjective refraction and Visual Acuity (VA)) and safety (tilt, decentration and posterior chamber opacification (PCO)) in a prospective series of 40 patients after bilateral implantation of AcrySof Natural ReSTOR (Model SN60D3) or AcrySof Natural Monofocal (Model SN60AT)
* to assess patient satisfaction before and after implant

ELIGIBILITY:
Inclusion:

* Written informed consent
* Age: ≥ 50 years ≤ 75 years
* Bilateral age related cataract, to be extracted and followed by the implantation of Posterior Chamber Intraocular Lenses (IOLs)
* Pre-operative and post-operative astigmatism ≤ 1 Diopter (D), as from Keratometry readings
* Potential post operative Visual Acuity (VA) ≥ 20/40
* Second eye surgery to take place no longer than 45 days after the first implant

Exclusion:

* Irregular optical aberrations;
* Pupil diameter in scotopic conditions more than 6 mm
* Degenerative visual pathologies (ex: Age-related Macular Degeneration (AMD))
* Other exclusions as from ReSTOR Directions for Use (DFU)

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2007-05; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Contact Alcon Call Center for Trial Locations, Fort Worth, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 35 patients, diagnosed with bilateral cataracts age related, requiring extraction of cataracts in both eyes followed by implantation of a posterior chamber intraocular lens, were recruited.
Pre-assignment Details: Patients meeting the inclusion/exclusion criteria were enrolled.
Groups:
- SN60D3: Intraocular Lens Acrysof Natural Restor SN60D3
- SN60AT: Intraocular Lens Acrysof Natural Monofocal SN60AT
Period: Overall Study
Arm/Group | SN60D3 | SN60AT
Started | 17 | 18
Completed | 16 | 15
Not Completed | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SN60D3 | SN60AT | Total
Number analyzed (Participants) | 17 | 18 | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 6 | 9
  >=65 years | 14 | 12 | 26
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 21
  Male | 7 | 7 | 14

OUTCOME MEASURES:

1. Primary Outcome: Near Best Corrected Visual Acuity (BCVA) - Binocular
Description: Percentage of patients with Near Visual Acuity (VA) ≥ 6.5/10 (≤ 0.18 LogMAR) at visit 8 (six months after implantation of the 2nd eye). This test was conducted binocularly and with best correction. The effect of treatment was tested by Chi-square test. VA is acuteness or clearness of vision, which is dependent on the sharpness of the retinal focus within the eye and the sensitivity of the interpretative faculty of the brain. VA is measured in logMAR which is the "logarithm of the minimum angle of resolution". A lower logMAR value indicates better VA.
Time Frame: 6 months after second eye implantation
Population: The # of subjects analyzed does not match the # of subjects in the participant flow as Near Visual Acuity (VA) was analyzed in the Intent To Treat population (N=16 for both groups). VA data were collected in different units (ie c, twentieth, decimal, Jaeger) & were converted to LogMAR after inclusion in the database leading to data approximations.
Measure: Number; unit: Percentage of Participants
Arm/Group | SN60D3 | SN60AT
Number analyzed (Participants) | 16 | 16
Percentage of Participants | 87.5 | 100

2. Primary Outcome: Near Uncorrected Visual Acuity (UCVA) Binocular
Description: Percentage of patients with Near Visual Acuity (VA) ≥ 6.5/10 (≤ 0.18 LogMAR) at visit 8 (six months after implantation of the 2nd eye). This test was conducted binocularly and with no correction. The effect of treatment was tested by Chi-square test. VA is acuteness or clearness of vision, which is dependent on the sharpness of the retinal focus within the eye and the sensitivity of the interpretative faculty of the brain. VA is measured in logMAR which is the "logarithm of the minimum angle of resolution". A lower logMAR value indicates better VA.
Time Frame: 6 months after second eye implantation
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | SN60D3 | SN60AT
Number analyzed (Participants) | 16 | 16
Percentage of Participants | 100 | 31.25

3. Primary Outcome: Near Best Corrected Visual Acuity Left Eye (BCVA LE)
Description: Percentage of patients with Near Visual Acuity (VA) ≥ 6.5/10 (≤ 0.18 LogMAR) at visit 8 (six months after implantation of the 2nd eye). This test was conducted monocularly (left eye only) and with best correction. The effect of treatment was tested by Chi-square test. VA is acuteness or clearness of vision, which is dependent on the sharpness of the retinal focus within the eye and the sensitivity of the interpretative faculty of the brain. VA is measured in logMAR which is the "logarithm of the minimum angle of resolution". A lower logMAR value indicates better VA.
Time Frame: 6 months after second eye implantation
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | SN60D3 | SN60AT
Number analyzed (Participants) | 16 | 16
Percentage of Participants | 87.5 | 100

4. Primary Outcome: Near Uncorrected Visual Acuity Left Eye (UCVA LE)
Description: Percentage of patients with Near Visual Acuity (VA) ≥ 6.5/10 (≤ 0.18 LogMAR) at visit 8 (six months after implantation of the 2nd eye). This test was conducted monocularly (left eye only) and with no correction. The effect of treatment was tested by Chi-square test. VA is acuteness or clearness of vision, which is dependent on the sharpness of the retinal focus within the eye and the sensitivity of the interpretative faculty of the brain. VA is measured in logMAR which is the "logarithm of the minimum angle of resolution". A lower logMAR value indicates better VA.
Time Frame: 6 months after second eye implantation
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | SN60D3 | SN60AT
Number analyzed (Participants) | 16 | 16
Percentage of Participants | 100 | 18.75

5. Primary Outcome: Near Best Corrected Visual Acuity Right Eye (BCVA RE)
Description: Percentage of patients with Near Visual Acuity (VA) ≥ 6.5/10 (≤ 0.18 LogMAR) at visit 8 (six months after implantation of the 2nd eye). This test was conducted monocularly (right eye only) and with best correction. The effect of treatment was tested by Chi-square test. VA is acuteness or clearness of vision, which is dependent on the sharpness of the retinal focus within the eye and the sensitivity of the interpretative faculty of the brain. VA is measured in logMAR which is the "logarithm of the minimum angle of resolution". A lower logMAR value indicates better VA.
Time Frame: 6 months after second eye implantation
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | SN60D3 | SN60AT
Number analyzed (Participants) | 16 | 16
Percentage of Participants | 68.75 | 100

6. Primary Outcome: Near Uncorrected Visual Acuity Right Eye (UCVA RE)
Description: Percentage of patients with Near Visual Acuity (VA) ≥ 6.5/10 (≤ 0.18 LogMAR) at visit 8 (six months after implantation of the 2nd eye). This test was conducted monocularly (right eye only) and with no correction. The effect of treatment was tested by Chi-square test. VA is acuteness or clearness of vision, which is dependent on the sharpness of the retinal focus within the eye and the sensitivity of the interpretative faculty of the brain. VA is measured in logMAR which is the "logarithm of the minimum angle of resolution". A lower logMAR value indicates better VA.
Time Frame: 6 months after second eye implantation
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | SN60D3 | SN60AT
Number analyzed (Participants) | 16 | 16
Percentage of Participants | 100 | 25

ADVERSE EVENTS:
Time Frame: Visit 2 (1st eye implant) through Visit 8 (6 months following 2nd implant)
Arm/Group | SN60D3 | SN60AT
Serious Adverse Events (participants affected / at risk) | 1/17 | 1/118
Other Adverse Events (participants affected / at risk) | 2/17 | 3/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | SN60D3 (N=17) | SN60AT (N=118)
Aortic aneurysm (Vascular disorders) | 1 (1) | 0/18 (0) — Not device related
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1/18 (1) — Not device related
OTHER ADVERSE EVENTS (reported when occurring in more than 1.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SN60D3 (N=17) | SN60AT (N=18)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
hernia hiatal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stenosis and insufficiency of lacrimal passages (Eye disorders) | 0 (0) | 1 (1)
Corneal membrane disorder NOS (Eye disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Visual acuity data were collected in different units (i.e. c, twentieth, decimal, Jaeger) and were converted to LogMAR after inclusion in the database. This led to inevitable approximations of the data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any formal presentation of data publication from this study has to be a joint presentation from both the Investigators and the Sponsor. Being the study multicentric, it is mandatory that the first publication is based on data from all the centres, analysed according to the protocol. Data from a single Centre can not be presented, unless there is a formal agreement from the other Investigators and Alcon.